CLINICAL TRIAL: NCT03934554
Title: ARS Experimentation Project: Improving Accessibility to the Renal Transplantation List
Brief Title: Improved Accessibility to the Renal Transplant List
Acronym: 2ALTR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Aider Montpellier : Dr Chalabi Lofti (Unknown); Aider Cèvennes et Confins Rhodaniens : Dr Mohajer Médérick (Unknown); Aider Nîmes : Philippe LAN YUE WAH (Unknown); Aider Lozère : Dr Hélène LERAY / Dr Cécile TURC-BARON (Unknown); Aider Perpignan : Dr Ahmed RACHI (Unknown); CHU de Nîmes : Pr Moranne Olivier (Unknown); CH de Perpignan : Dr Vela Carlos (Unknown); Centre d'Hémodialyse St Guilhem : Dr Argilès Angèl (Unknown); Clinique Médipôle Perpignan : Dr DECOURT Alexandre (Unknown); Clinique de Narbonne : Dr De Cornélissen François (Unknown); GCS Help : Dr Maria Eugenia Noguera Gonzales (Unknown); NephroCare Castelnau / Mas du Rochet / Lunel : Dr Basel Olivia (Unknown); NephroCare Béziers : Dr Baron Emmanuel (Unknown); NephroCare Nîmes / Bagnols : Dr Rousseau Philippe (Unknown); Villeneuve les Béziers : Dr Baron Emmanuel (Unknown); GCS eSanté : Sylvain Collet (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0138
Record Dates: First submitted 2019-04-25; First posted 2019-05-02 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Chronic End Stage Renal Failure
Keywords: Nephrology; Kidney transplant; Registration; Transplant waiting list

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Two 9 mL EDTA (ethylenediaminetetraacetic acid) blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In 2014, the "States General of Kidney" have allowed to assess the situation concerning the management of chronic kidney disease on the national territory. Ex-Languedoc-Roussillon has emerged as one of the French regions with a high dialysis / transplant ratio compared to other regions. Disparities in accessibility to the kidney transplant list were also very important. In the ex-Languedoc-Roussillon Region, the number of patients on the renal transplant list was lower than the national average (18.9 vs. 24.1%, respectively, according to the REIN 2015 report).

In 2015, the Regional Health Agency (ARS) ex-Languedoc-Roussillon, has published proposals to improve the healthcare of the patient in chronic end stage renal failure, and accessibility to the national waiting list for renal transplantation (CRISTAL).

To increase accessibility to the national waiting list for renal transplantation by improving the patient's healthcare, our project is based on the creation of a reinforced exchanges connexion between the hospital's nephrology services professionals, dialysis units and liberal nephrologists. This will include having regular meetings between dialysis nephrologists and CHU nephrologists. The proposals for this project were:

1. to organize multidisciplinary consultation meetings between transplant and dialysis professionals
2. to set up an exchange platform and communication tools built on the model of telemedicine (COVOTEM), common to the nephrology departments of the University Hospital Center, dialysis units.

This new device for the management of chronic end stage renal failure should increase the number of patients on the national renal transplantation waiting list. It should also make it possible to reduce the time between: firstly, the sending of the pre-registration file to the transplantation at Montpellier University Hospital and registration, and secondly between dialysis and registration.on waiting list.

The investigators hope that this experiment will increase the number of registrations on the National Kidney Transplantation Waitlist (CRISTAL). The implementation of this innovative tool should facilitate communication between nephrologists dialysis centers and nephrologists of CHU Montpellier, and accelerate the process of registration on the National Kidney Transplantation Waitlist.

If this platform proves to be easy to use and if the project's evaluation criteria show significant results, the platform could then be used to monitor patients in post-transplantation. Indeed, the data of patients who perform an alternating follow-up would be available for the referring nephrologists and for the transplant center. The further development of the platform would allow to create a mode of communication via this platform.

DETAILED DESCRIPTION:
Main Objective: Evolution of the number of patients, dialysed or not dialysed in the ex-Languedoc-Roussillon Region, acceding during the year, to a pre-transplant assessment for a registration on the national renal transplantation waiting list ( CRISTAL).

Secondary Objectives:

* Evolution of patient waiting times for registration on the national renal transplantation waiting list (CRISTAL)
* For incident cases: Evolution of the time between dialysis, and the date of registration on the transplant waiting list or the date of decision of temporary or definitive contraindication by nephrologists CHU Montpellier .
* Evolution of the delays between the date of reception of the pre-registration file by the nephrology department of the University Hospital and the closing date of the file (either a definitive inscription, a definitive contraindication or a temporary contraindication > 4 months)
* Evolution of the number of multidisciplinary consultation meetings performed without videoconferencing and videoconferencing between the dialysis center and Montpellier University Hospital
* Evaluation of exchanges between professionals involved in the course of care of the patient in chronic end stage renal failure

ELIGIBILITY:
Inclusion Criteria:

* Dialysis or non-dialysis patients with chronic renal insufficiency with a GFR < 20ml / min eligible for transplant
* Patient wishing to start the registration process at the transplant
* Patient giving consent for the transmission of his data via an electronic platform

Exclusion Criteria:

* Patient already enrolled
* Patient having a pathology with a life expectancy of less than two years
* Patient with serious psychiatric disorders , or dementia.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients dialysed or not dialysed with end stage renal failure, eligible for a pre-transplant assessment
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of patient dialysed or not dialysed acceding to a pre-transplant assessment for a registration on the national renal transplantation waiting list ( CRISTAL). | 1 year, up to the end of study
  Number of patient dialysed or not dialysed acceding to a pre-transplant assessment for a registration on the national renal transplantation waiting list ( CRISTAL).

SECONDARY OUTCOMES:
Number of files received by the nephrology department of Montpellier University Hospital on the COVOTEM platform | 1 year, up to the end of study
  Number of files received by the nephrology department of Montpellier University Hospital on the COVOTEM platform
Number of dialysis patients who had a pre-transplant evaluation | 1 year, up to the end of study
  Number of dialysis patients who had a pre-transplant evaluation
Number of non-dialysis patients who had a pre-transplant evaluation | 1 year, up to the end of study
  Number of non-dialysis patients who had a pre-transplant evaluation
Number of patients on temporary or definitive contraindications | 1 year, up to the end of study
  Number of patients on temporary or definitive contraindications
Average period between the dialysis of the patient and the reception of the pre-registration file by the nephrology department of Montpellier University Hospital | 1 year, up to the end of study
  Average period between the dialysis of the patient and the reception of the pre-registration file by the nephrology department of Montpellier University Hospital
Average period between the reception of the pre-registration file by the nephrology department of the University Hospital of Montpellier and the consultation appointment for registration | 1 year, up to the end of study
  Average period between the reception of the pre-registration file by the nephrology department of the University Hospital of Montpellier and the consultation appointment for registration
Average period between the reception of the pre-registration file | 1 year, up to the end of study
  Average period between the reception of the pre-registration file by the nephrology department of the CHU of Montpellier and the closing of the file (either a definitive inscription, a definitive contraindication, or a temporary contraindication > 4months)
Rate of participation of the centers in the experimentation (Number of files received by the nephrology department of the University Hospital Center of Montpellier per center) | 1 year, up to the end of study
  Rate of participation of the centers in the experimentation (Number of files received by the nephrology department of the University Hospital Center of Montpellier per center)
Number of multidisciplinary consultation meetings performed without videoconferencing or videoconferencing between the dialysis center and Montpellier University Hospital Center | 1 year, up to the end of study
  Number of multidisciplinary consultation meetings performed without videoconferencing or videoconferencing between the dialysis center and Montpellier University Hospital Center
Average period between the consultation appointment and the closing of the file (either a definitive inscription, a definitive contraindication, or a temporary contraindication > 4months | 1 year, up to the end of study
  Average period between the consultation appointment and the closing of the file (either a definitive inscription, a definitive contraindication, or a temporary contraindication > 4months
Number of non-dialysis patients with renal insufficiency enrolled preemptively on the national renal transplantation waiting list | 1 year, up to the end of study
  Number of non-dialysis patients with renal insufficiency enrolled preemptively on the national renal transplantation waiting list

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie DELMAS, Doctor, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC